CLINICAL TRIAL: NCT05384457
Title: The Breathe-(H)IT Trial: Multimodal High Intensity Training to Improve Diaphragm Functioning in Persons With Chronic Nonspecific Low Back Pain
Brief Title: High Intensity Training to Improve Diaphragm Functioning in Persons With Chronic Nonspecific Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hasselt University (Other)
Collaborators: KU Leuven (Other); Maastricht University (Other)
Responsible Party: Principal Investigator, Annick Timmermans, Prof. Dr., Hasselt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B1152021000029
Record Dates: First submitted 2022-05-11; First posted 2022-05-20 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Low Back Pain; Chronic Low-back Pain; Chronic Pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High intensity training (HIT) (Experimental): Each participant will follow 24 therapy sessions (2 x 1.5 hours/week). The experimental group will perform a multimodal HIT protocol. Cardiorespiratory training will consist of a high-intensity interval training protocol on a cycle ergometer. After a five-minute warm-up, interval training will start, consisting of five one-minute bouts (110 RPM at 100% VO2max workload), separated by one minute of active rest (75 RPM at 50% VO2max workload). Limb strength training will consist of a circuit of three upper-body (vertical traction, chest press, arm curl) and three lower-body exercises (leg curl, leg press, leg extension) executed at 80% of the one repetition maximum. Core muscle training will consist of a circuit of six static core exercises (glute bridge, glute clam, superman back extension, adapted plank, adapted side plank, shoulder retraction with hip hinge) at 60% of the maximal voluntary contraction.
  Interventions: Other: High intensity training
- Moderate intensity training (MIT) (Active Comparator): Each participant will follow 24 therapy sessions (2 x 1.5 hours/week). The control group will perform a multimodal MIT protocol. Cardiorespiratory training will consist of a moderate-intensity continuous training protocol on a cycle ergometer. After a five-minute warm up, participants start continuous training comprising of 14 minutes of moderate-intensity cycling (90RPM at 60%VO2max workload). The duration will increase weekly with 1'40'' up to 22'40''. Limb strength training will consist of a circuit of three upper-body (vertical traction, chest press, arm curl) and three lower-body exercises (leg curl, leg press, leg extension) executed at 60% of the one repetition maximum. Core muscle training will be identical to the protocol described in 'Core muscle training HIT' with the exception of the exercise intensity. Only exercises with low relative core muscle activation will be used.
  Interventions: Other: Moderate intensity training

INTERVENTIONS:
Other: High intensity training — Participants will follow an exercise therapy program consisting of cardiorespiratory training, limb strength training and core muscle training.
  Arms: High intensity training (HIT)
Other: Moderate intensity training — Participants will follow an exercise therapy program consisting of cardiorespiratory training, limb strength training and core muscle training.
  Arms: Moderate intensity training (MIT)

SUMMARY:
This randomized controlled trial aims to investigate 1) the effects of high intensity training (HIT) compared to moderate intensity training (MIT) on diaphragm muscle strength, -endurance, -fatigue and -activation, 2) to which extent these changes in diaphragm functioning are related to changes in cardiorespiratory fitness, postural control, pain and disability after HIT versus MIT, 3) to which extent depressive mood and anxiety moderate the effects of HIT on diaphragm functioning in persons with chronic nonspecific low back pain (CNSLBP). The investigators hypothize that HIT improves diaphragm functioning more compared to MIT in persons with CNSLBP.

DETAILED DESCRIPTION:
Low back pain is the number one cause of disability worldwide with important socio-economic implications. In Belgium, 7 out of 10 persons will suffer from low back pain during their life, and 29% of all sick leave days are due to it. Chronic low back pain is defined as persistent pain for a period of minimal 12 weeks. In 85-90% of the CLBP cases, the pain cannot be attributed to a definitive underlying pathoanatomical cause, and is therefore labelled as chronic nonspecific low back pain (CNSLBP).

International guidelines recommend exercise therapy as the first-choice treatment for CNSLBP. A crucial factor within this context is exercise intensity. Indeed, multimodal high intensity training (HIT) leads to higher improvements in disability and cardiorespiratory fitness compared to moderate intensity training (MIT) in persons with CNSLBP. However, the underlying mechanisms for the additional value of a HIT approach remain largely unknown. Interestingly, low back pain is associated with impairments in diaphragm function, as the diaphragm is not only a principal inspiratory muscle, but also plays an essential role in postural control. The latter is a key factor in the development and maintenance of CNSLBP.

In this randomized controlled trial, 64 persons with CNSLBP will be recruited through local distribution of flyers and adverts on social media. The sample size calculation is based on (1) the therapeutic effects of a 12-week HIT program (compared to a MIT program) on the maximal oxygen uptake (VO2max) in persons with CNSLBP and (2) the therapeutic effects of a 8-week high-intensity inspiratory muscle training program (compared to a low-intensity inspiratory muscle training program) on the maximal inspiratory pressure (MIP) in persons with CNSLBP. These outcomes were chosen as they relate to the respiratory system and are thus most fitting to indicate possible effects on diaphragm functioning. The sample size calculation is based on the requirement of a minimal clinically important difference of 3-3.5ml/kg/min (VO2max) and 17.2 H2O (MIP). The power calculation resulted in a total of 63 persons. Therefore, the investigators plan to recruit 64 patients.

Participants will be randomly assigned to a HIT program or a MIT program. Primary outcomes are diaphragm muscle strength, -endurance, -fatigue and - activation. Secondary outcomes are cardiorespiratory fitness, postural control, pain, disability, depressive mood and anxiety. Primary and secondary outcomes will be assessed at 5 timepoints (0 weeks, 6 weeks, 12 weeks, 3 months after intervention, 12 months after intervention).

To analyze the data, JMP Pro (15.2 SAS Institute Inc, Cary, USA) will be used. Descriptive statistics will be used to display baseline group characteristics. To evaluate between-group differences (i.e. the effectiveness of the HIT vs MIT intervention), a linear mixed model will be fitted with 'time' and 'group' as covariates, and incorporated random intercepts for the participants to account for the within-subject variation. To evaluate associations between diaphragm functioning and predictors/mediators for therapy success, correlations and multivariate regression analysis will be used.

ELIGIBILITY:
Inclusion Criterian (CNSLBP patients):

* Dutch-speaking
* Adults (age 18-65 years)
* Chronic low back pain (i.e. pain localized below the costal margin and above the inferior gluteal folds, with or without referred leg pain for a period of at least twelve weeks), with a non-specific origin (i.e. pain of a nociceptive mechanical nature, not attributable to a recognizable, known, specific pathology, e.g. infection, tumour, osteoporosis, fracture, structural deformity, inflammatory disorder, radicular syndrome, or cauda equina syndrome)

Exclusion Criteria (CNSLBP patients):

* History of spinal fusion
* A musculoskeletal disorder aside from chronic nonspecific low back pain that could affect the correct execution of the therapy program
* Baseline characteristics that could affect the evaluation of the outcomes (a pacemaker, a chronic obstructive respiratory disorder, or known balance/vestibular problems)
* Severe comorbidities (e.g., paresis or sensory disturbances of neurological origin, diabetes mellitus, rheumatoid arthritis)
* Ongoing compensation claims
* Negative advice from the general practitioner regarding sports medical screening
* Pregnancy
* Persons that are not able to attend regular appointments

Inclusion Criteria (healthy volunteers):

* Dutch-speaking
* Adults (age 18-65 years)
* No acute or chronic complaints

Exclusion Criteria (healthy volunteers):

* History of spinal fusion
* Baseline characteristics that could affect the evaluation of the outcomes (a pacemaker, a chronic obstructive respiratory disorder, or known balance/vestibular problems)
* Severe comorbidities (e.g., paresis or sensory disturbances of neurological origin, diabetes mellitus, rheumatoid arthritis)
* Ongoing compensation claims
* Negative advice from the general practitioner regarding sports medical screening
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-08-22 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Diaphragm strength | PRE (baseline)
  Maximal inspiratory pressure (MIP) is a reliable measure to quantify inspiratory muscle strength. MIP will be measured at residual volume according to the method of Black and Hyatt using an electronic pressure transducer (POWERbreathe International Ltd., type KH2, Warwickshire, UK). A minimum of five repetitions will be performed, and tests will be repeated until there is less than 5% difference between the best and second-best test. The highest pressure sustained over 1 s will be defined as MIP, and compared with reference values.
Diaphragm strength | MID (6 weeks)
  Maximal inspiratory pressure (MIP) is a reliable measure to quantify inspiratory muscle strength. MIP will be measured at residual volume according to the method of Black and Hyatt using an electronic pressure transducer (POWERbreathe International Ltd., type KH2, Warwickshire, UK). A minimum of five repetitions will be performed, and tests will be repeated until there is less than 5% difference between the best and second-best test. The highest pressure sustained over 1 s will be defined as MIP.
Diaphragm strength | POST (12 weeks)
  Maximal inspiratory pressure (MIP) is a reliable measure to quantify inspiratory muscle strength. MIP will be measured at residual volume according to the method of Black and Hyatt using an electronic pressure transducer (POWERbreathe International Ltd., type KH2, Warwickshire, UK). A minimum of five repetitions will be performed, and tests will be repeated until there is less than 5% difference between the best and second-best test. The highest pressure sustained over 1 s will be defined as MIP.
Diaphragm strength | FU1 (3 months follow-up)
  Maximal inspiratory pressure (MIP) is a reliable measure to quantify inspiratory muscle strength. MIP will be measured at residual volume according to the method of Black and Hyatt using an electronic pressure transducer (POWERbreathe International Ltd., type KH2, Warwickshire, UK). A minimum of five repetitions will be performed, and tests will be repeated until there is less than 5% difference between the best and second-best test. The highest pressure sustained over 1 s will be defined as MIP.
Diaphragm strength | FU2 (12 months follow-up)
  Maximal inspiratory pressure (MIP) is a reliable measure to quantify inspiratory muscle strength. MIP will be measured at residual volume according to the method of Black and Hyatt using an electronic pressure transducer (POWERbreathe International Ltd., type KH2, Warwickshire, UK). A minimum of five repetitions will be performed, and tests will be repeated until there is less than 5% difference between the best and second-best test. The highest pressure sustained over 1 s will be defined as MIP.
Diaphragm endurance | PRE (baseline)
  Participants will undergo an inspiratory resistive loading protocol at a fixed intensity of 80% of MIP (POWERbreathe International Ltd., type KH2, Warwickshire, UK). The participants will be instructed to inhale maximally and as rapidly as possible at a frequency of 15 breaths/minute and a 0.5 duty cycle. The time to task failure will be recorded as the inspiratory muscle endurance time.
Diaphragm endurance | POST (12 weeks)
  Participants will undergo an inspiratory resistive loading protocol at a fixed intensity of 80% of MIP (POWERbreathe International Ltd., type KH2, Warwickshire, UK). The participants will be instructed to inhale maximally and as rapidly as possible at a frequency of 15 breaths/minute and a 0.5 duty cycle. The time to task failure will be recorded as the inspiratory muscle endurance time.
Diaphragm fatigue | PRE (baseline)
  Diaphragm fatigue is defined as a reduction in the ability to produce force/pressure following contractile activity. First, MIP will be measured using an electronic pressure transducer (POWERbreathe International Ltd., type KH2, Warwickshire, UK). Then, the participant will perform a maximal cardiopulmonary exercise test (CPET). After the CPET, the MIP-measurement will be repeated. The difference between the MIP before and after the CPET will be used as a measure of diaphragm fatigue.
Diaphragm fatigue | MID (6 weeks)
  Diaphragm fatigue is defined as a reduction in the ability to produce force/pressure following contractile activity. First, MIP will be measured using an electronic pressure transducer ((POWERbreathe International Ltd., type KH2, Warwickshire, UK). Then, the participant will perform a maximal cardiopulmonary exercise test (CPET). After the CPET, the MIP-measurement will be repeated. The difference between the MIP before and after the CPET will be used as a measure of diaphragm fatigue.
Diaphragm fatigue | POST (12 weeks)
  Diaphragm fatigue is defined as a reduction in the ability to produce force/pressure following contractile activity. First, MIP will be measured using an electronic pressure transducer (POWERbreathe International Ltd., type KH2, Warwickshire, UK). Then, the participant will perform a maximal cardiopulmonary exercise test (CPET). After the CPET, the MIP-measurement will be repeated. The difference between the MIP before and after the CPET will be used as a measure of diaphragm fatigue.
Diaphragm fatigue | FU1 (3 months follow-up)
  Diaphragm fatigue is defined as a reduction in the ability to produce force/pressure following contractile activity. First, MIP will be measured using an electronic pressure transducer (POWERbreathe International Ltd., type KH2, Warwickshire, UK). Then, the participant will perform a maximal cardiopulmonary exercise test (CPET). After the CPET, the MIP-measurement will be repeated. The difference between the MIP before and after the CPET will be used as a measure of diaphragm fatigue.
Diaphragm fatigue | FU2 (12 months follow-up)
  Diaphragm fatigue is defined as a reduction in the ability to produce force/pressure following contractile activity. First, MIP will be measured using an electronic pressure transducer (POWERbreathe International Ltd., type KH2, Warwickshire, UK). Then, the participant will perform a maximal cardiopulmonary exercise test (CPET). After the CPET, the MIP-measurement will be repeated. The difference between the MIP before and after the CPET will be used as a measure of diaphragm fatigue.
Diaphragm activation (amplitude) | PRE (baseline)
  Diaphragm activation will be measured in terms of electromyography (EMG) amplitude. Surface EMG will be acquired throughout the postural control tasks and cardiopulmonary exercise test to measure muscle activation from the costal diaphragm/intercostals, scalene, parasternal intercostal, and sternocleidomastoid.
Diaphragm activation (amplitude) | MID (6 weeks)
  Diaphragm activation will be measured in terms of electromyography (EMG) amplitude. Surface EMG will be acquired throughout the postural control tasks and cardiopulmonary exercise test to measure muscle activation from the costal diaphragm/intercostals, scalene, parasternal intercostal, and sternocleidomastoid.
Diaphragm activation (amplitude) | POST (12 weeks)
  Diaphragm activation will be measured in terms of electromyography (EMG) amplitude. Surface EMG will be acquired throughout the postural control tasks and cardiopulmonary exercise test to measure muscle activation from the costal diaphragm/intercostals, scalene, parasternal intercostal, and sternocleidomastoid.
Diaphragm activation (amplitude) | FU1 (3 months follow-up)
  Diaphragm activation will be measured in terms of electromyography (EMG) amplitude. Surface EMG will be acquired throughout the postural control tasks and cardiopulmonary exercise test to measure muscle activation from the costal diaphragm/intercostals, scalene, parasternal intercostal, and sternocleidomastoid.
Diaphragm activation (amplitude) | FU2 (12 months follow-up)
  Diaphragm activation will be measured in terms of electromyography (EMG) amplitude. Surface EMG will be acquired throughout the postural control tasks and cardiopulmonary exercise test to measure muscle activation from the costal diaphragm/intercostals, scalene, parasternal intercostal, and sternocleidomastoid.
Diaphragm activation (timing) | PRE (baseline)
  Diaphragm activation will be measured in terms of electromyography (EMG) timing. Surface EMG will be acquired throughout the postural control tasks and cardiopulmonary exercise test to measure muscle activation from the costal diaphragm/intercostals, scalene, parasternal intercostal, and sternocleidomastoid.
Diaphragm activation (timing) | MID (6 weeks)
  Diaphragm activation will be measured in terms of electromyography (EMG) timing. Surface EMG will be acquired throughout the postural control tasks and cardiopulmonary exercise test to measure muscle activation from the costal diaphragm/intercostals, scalene, parasternal intercostal, and sternocleidomastoid.
Diaphragm activation (timing) | POST (12 weeks)
  Diaphragm activation will be measured in terms of electromyography (EMG) timing. Surface EMG will be acquired throughout the postural control tasks and cardiopulmonary exercise test to measure muscle activation from the costal diaphragm/intercostals, scalene, parasternal intercostal, and sternocleidomastoid.
Diaphragm activation (timing) | FU1 (3 months follow-up)
  Diaphragm activation will be measured in terms of electromyography (EMG) timing. Surface EMG will be acquired throughout the postural control tasks and cardiopulmonary exercise test to measure muscle activation from the costal diaphragm/intercostals, scalene, parasternal intercostal, and sternocleidomastoid.
Diaphragm activation (timing) | FU2 (12 months follow-up)
  Diaphragm activation will be measured in terms of electromyography (EMG) timing. Surface EMG will be acquired throughout the postural control tasks and cardiopulmonary exercise test to measure muscle activation from the costal diaphragm/intercostals, scalene, parasternal intercostal, and sternocleidomastoid.

SECONDARY OUTCOMES:
Modified Oswestry Disability Index (MODI) | PRE (baseline)
  The Modified Oswestry Disability Index is a valid and reliable questionnaire for evaluating constraints experienced by people in their daily activities due to chronic low back pain. It consists of ten items scored on a five-point scale. The total score is expressed in percentage (min. 0%, max. 100%) and displays the degree of functional limitation. A higher score indicates a higher degree of functional limitation.
Modified Oswestry Disability Index (MODI) | MID (6 weeks)
  The Modified Oswestry Disability Index is a valid and reliable questionnaire for evaluating constraints experienced by people in their daily activities due to chronic low back pain. It consists of ten items scored on a five-point scale. The total score is expressed in percentage (min. 0%, max. 100%) and displays the degree of functional limitation. A higher score indicates a higher degree of functional limitation.
Modified Oswestry Disability Index (MODI) | POST (12 weeks)
  The Modified Oswestry Disability Index is a valid and reliable questionnaire for evaluating constraints experienced by people in their daily activities due to chronic low back pain. It consists of ten items scored on a five-point scale. The total score is expressed in percentage (min. 0%, max. 100%) and displays the degree of functional limitation. A higher score indicates a higher degree of functional limitation.
Modified Oswestry Disability Index (MODI) | FU1 (3 months follow-up)
  The Modified Oswestry Disability Index is a valid and reliable questionnaire for evaluating constraints experienced by people in their daily activities due to chronic low back pain. It consists of ten items scored on a five-point scale. The total score is expressed in percentage (min. 0%, max. 100%) and displays the degree of functional limitation. A higher score indicates a higher degree of functional limitation.
Modified Oswestry Disability Index (MODI) | FU2 (12 months follow-up)
  The Modified Oswestry Disability Index is a valid and reliable questionnaire for evaluating constraints experienced by people in their daily activities due to chronic low back pain. It consists of ten items scored on a five-point scale. The total score is expressed in percentage (min. 0%, max. 100%) and displays the degree of functional limitation. A higher score indicates a higher degree of functional limitation.
Brief Pain Inventory (BPI) | PRE (baseline)
  The Brief Pain Inventory assesses the severity of pain, its impact on functioning, the location of pain, pain medications, and the amount of pain relief in the past 24 hours. The body chart of this questionnaire will be used to record the extent of pain, using the pain drawing method. The extent of pain might indicate the presence of widespread pain, which has been associated with altered nociceptive pain processing in chronic joint pain. The BPI scale defines pain as follows:
  * Worst Pain Score: 1 - 4 = Mild Pain
  * Worst Pain Score: 5 - 6 = Moderate Pain
  * Worst Pain Score: 7 - 10 = Severe Pain
Brief Pain Inventory (BPI) | MID (6 weeks)
  The Brief Pain Inventory assesses the severity of pain, its impact on functioning, the location of pain, pain medications, and the amount of pain relief in the past 24 hours. The body chart of this questionnaire will be used to record the extent of pain, using the pain drawing method. The extent of pain might indicate the presence of widespread pain, which has been associated with altered nociceptive pain processing in chronic joint pain. The BPI scale defines pain as follows:
  * Worst Pain Score: 1 - 4 = Mild Pain
  * Worst Pain Score: 5 - 6 = Moderate Pain
  * Worst Pain Score: 7 - 10 = Severe Pain
Brief Pain Inventory (BPI) | POST (12 weeks)
  The Brief Pain Inventory assesses the severity of pain, its impact on functioning, the location of pain, pain medications, and the amount of pain relief in the past 24 hours. The body chart of this questionnaire will be used to record the extent of pain, using the pain drawing method. The extent of pain might indicate the presence of widespread pain, which has been associated with altered nociceptive pain processing in chronic joint pain. The BPI scale defines pain as follows:
  * Worst Pain Score: 1 - 4 = Mild Pain
  * Worst Pain Score: 5 - 6 = Moderate Pain
  * Worst Pain Score: 7 - 10 = Severe Pain
Brief Pain Inventory (BPI) | FU1 (3 months follow-up)
  The Brief Pain Inventory assesses the severity of pain, its impact on functioning, the location of pain, pain medications, and the amount of pain relief in the past 24 hours. The body chart of this questionnaire will be used to record the extent of pain, using the pain drawing method. The extent of pain might indicate the presence of widespread pain, which has been associated with altered nociceptive pain processing in chronic joint pain. The BPI scale defines pain as follows:
  * Worst Pain Score: 1 - 4 = Mild Pain
  * Worst Pain Score: 5 - 6 = Moderate Pain
  * Worst Pain Score: 7 - 10 = Severe Pain
Brief Pain Inventory (BPI) | FU2 (12 months follow-up)
  The Brief Pain Inventory assesses the severity of pain, its impact on functioning, the location of pain, pain medications, and the amount of pain relief in the past 24 hours. The body chart of this questionnaire will be used to record the extent of pain, using the pain drawing method. The extent of pain might indicate the presence of widespread pain, which has been associated with altered nociceptive pain processing in chronic joint pain. The BPI scale defines pain as follows:
  * Worst Pain Score: 1 - 4 = Mild Pain
  * Worst Pain Score: 5 - 6 = Moderate Pain
  * Worst Pain Score: 7 - 10 = Severe Pain
Beck Depression Inventory (BDI) | PRE (baseline)
  The Beck Depression Inventory is widely used as a self-reported questionnaire for assessing depression in patients with chronic pain. It consists of 21 items scored on a four-point scale (0-3). Item scores are summed to obtain the total score, with a higher total score indicating greater depression.
Beck Depression Inventory (BDI) | POST (12 weeks)
  The Beck Depression Inventory is widely used as a self-reported questionnaire for assessing depression in patients with chronic pain. It consists of 21 items scored on a four-point scale (0-3). Item scores are summed to obtain the total score, with a higher total score indicating greater depression.
Beck Depression Inventory (BDI) | FU2 (12 months follow-up)
  The Beck Depression Inventory is widely used as a self-reported questionnaire for assessing depression in patients with chronic pain. It consists of 21 items scored on a four-point scale (0-3). Item scores are summed to obtain the total score, with a higher total score indicating greater depression.
State-Trait Anxiety Inventory (STAI) | PRE (baseline)
  The State-Trait Anxiety Inventory is a questionnaire for assessing state anxiety (i.e. anxiety about an event) and trait anxiety (i.e. anxiety as a personal characteristic). It consists of 40 items scored on a four-point scale. Item scores are added to obtain the total score. The score of the STAI varies from a minimum score of 20 to a maximum score of 80 on both the STAI-state and STAI-trait subscales. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
State-Trait Anxiety Inventory (STAI) | POST (12 weeks)
  The State-Trait Anxiety Inventory is a questionnaire for assessing state anxiety (i.e. anxiety about an event) and trait anxiety (i.e. anxiety as a personal characteristic). It consists of 40 items scored on a four-point scale. Item scores are added to obtain the total score. The score of the STAI varies from a minimum score of 20 to a maximum score of 80 on both the STAI-state and STAI-trait subscales. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
State-Trait Anxiety Inventory (STAI) | FU2 (12 months follow-up)
  The State-Trait Anxiety Inventory is a questionnaire for assessing state anxiety (i.e. anxiety about an event) and trait anxiety (i.e. anxiety as a personal characteristic). It consists of 40 items scored on a four-point scale. Item scores are added to obtain the total score. The score of the STAI varies from a minimum score of 20 to a maximum score of 80 on both the STAI-state and STAI-trait subscales. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80).
Relative proprioceptive weighting ratio | PRE (baseline)
  A force plate will measure center of pressure (COP) displacement in response to ankle and lumbar muscle vibration during upright standing. If a person relies on proprioception from the vibrated muscle, an illusion of loss of balance will occur. To compensate, participants will move their COP in the opposite direction. When the triceps surae muscles are vibrated, a postural sway in a backward direction is expected, whereas during lumbar paraspinal muscle vibration, a forward postural body sway is expected. The amount of COP displacement during local vibration may represent the extent to which a person makes use of the proprioceptive signals of the vibrated muscles to maintain the upright posture. Reliance on ankle vs. lumbar proprioception will be calculated as the Relative Proprioceptive Weighting (RPW) ratio: RPW= AbsAnkle/(AbsAnkle + AbsLumbar). 'AbsAnkle' and 'AbsLumbar' refer to the absolute COP displacement during ankle and lumbar muscle vibration, respectively.
Relative proprioceptive weighting ratio | MID (6 weeks)
  A force plate will measure center of pressure (COP) displacement in response to ankle and lumbar muscle vibration during upright standing. If a person relies on proprioception from the vibrated muscle, an illusion of loss of balance will occur. To compensate, participants will move their COP in the opposite direction. When the triceps surae muscles are vibrated, a postural sway in a backward direction is expected, whereas during lumbar paraspinal muscle vibration, a forward postural body sway is expected. The amount of COP displacement during local vibration may represent the extent to which a person makes use of the proprioceptive signals of the vibrated muscles to maintain the upright posture. Reliance on ankle vs. lumbar proprioception will be calculated as the Relative Proprioceptive Weighting (RPW) ratio: RPW= AbsAnkle/(AbsAnkle + AbsLumbar). 'AbsAnkle' and 'AbsLumbar' refer to the absolute COP displacement during ankle and lumbar muscle vibration, respectively.
Relative proprioceptive weighting ratio | POST (12 weeks)
  A force plate will measure center of pressure (COP) displacement in response to ankle and lumbar muscle vibration during upright standing. If a person relies on proprioception from the vibrated muscle, an illusion of loss of balance will occur. To compensate, participants will move their COP in the opposite direction. When the triceps surae muscles are vibrated, a postural sway in a backward direction is expected, whereas during lumbar paraspinal muscle vibration, a forward postural body sway is expected. The amount of COP displacement during local vibration may represent the extent to which a person makes use of the proprioceptive signals of the vibrated muscles to maintain the upright posture. Reliance on ankle vs. lumbar proprioception will be calculated as the Relative Proprioceptive Weighting (RPW) ratio: RPW= AbsAnkle/(AbsAnkle + AbsLumbar). 'AbsAnkle' and 'AbsLumbar' refer to the absolute COP displacement during ankle and lumbar muscle vibration, respectively.
Relative proprioceptive weighting ratio | FU1 (3 months follow-up)
  A force plate will measure center of pressure (COP) displacement in response to ankle and lumbar muscle vibration during upright standing. If a person relies on proprioception from the vibrated muscle, an illusion of loss of balance will occur. To compensate, participants will move their COP in the opposite direction. When the triceps surae muscles are vibrated, a postural sway in a backward direction is expected, whereas during lumbar paraspinal muscle vibration, a forward postural body sway is expected. The amount of COP displacement during local vibration may represent the extent to which a person makes use of the proprioceptive signals of the vibrated muscles to maintain the upright posture. Reliance on ankle vs. lumbar proprioception will be calculated as the Relative Proprioceptive Weighting (RPW) ratio: RPW= AbsAnkle/(AbsAnkle + AbsLumbar). 'AbsAnkle' and 'AbsLumbar' refer to the absolute COP displacement during ankle and lumbar muscle vibration, respectively.
Relative proprioceptive weighting ratio | FU2 (12 months follow-up)
  A force plate will measure center of pressure (COP) displacement in response to ankle and lumbar muscle vibration during upright standing. If a person relies on proprioception from the vibrated muscle, an illusion of loss of balance will occur. To compensate, participants will move their COP in the opposite direction. When the triceps surae muscles are vibrated, a postural sway in a backward direction is expected, whereas during lumbar paraspinal muscle vibration, a forward postural body sway is expected. The amount of COP displacement during local vibration may represent the extent to which a person makes use of the proprioceptive signals of the vibrated muscles to maintain the upright posture. Reliance on ankle vs. lumbar proprioception will be calculated as the Relative Proprioceptive Weighting (RPW) ratio: RPW= AbsAnkle/(AbsAnkle + AbsLumbar). 'AbsAnkle' and 'AbsLumbar' refer to the absolute COP displacement during ankle and lumbar muscle vibration, respectively.
Thermal Detection and Pain Threshold Temperatures | PRE (baseline)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc Advanced Thermosensory Stimulator (TSA) - 2 system will be used to perform a standardized test protocol.
  Detection and pain threshold temperatures (in °C) will be assessed locally (at the most painful site of the lower back) and remotely (at the contralateral wrist) using the TSA limits protocol:
  * Cold Detection Threshold (CDT)
  * Warmth Detection Threshold (WDT)
  * Cold Pain Threshold (CPT)
  * Heat Pain Threshold (HPT)
Thermal Detection and Pain Threshold Temperatures | MID (6 weeks)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc Advanced Thermosensory Stimulator (TSA) - 2 system will be used to perform a standardized test protocol.
  Detection and pain threshold temperatures (in °C) will be assessed locally (at the most painful site of the lower back) and remotely (at the contralateral wrist) using the TSA limits protocol:
  * Cold Detection Threshold (CDT)
  * Warmth Detection Threshold (WDT)
  * Cold Pain Threshold (CPT)
  * Heat Pain Threshold (HPT)
Thermal Detection and Pain Threshold Temperatures | POST (12 weeks)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc Advanced Thermosensory Stimulator (TSA) - 2 system will be used to perform a standardized test protocol.
  Detection and pain threshold temperatures (in °C) will be assessed locally (at the most painful site of the lower back) and remotely (at the contralateral wrist) using the TSA limits protocol:
  * Cold Detection Threshold (CDT)
  * Warmth Detection Threshold (WDT)
  * Cold Pain Threshold (CPT)
  * Heat Pain Threshold (HPT)
Thermal Detection and Pain Threshold Temperatures | FU1 (3 months follow-up)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc Advanced Thermosensory Stimulator (TSA) - 2 system will be used to perform a standardized test protocol.
  Detection and pain threshold temperatures (in °C) will be assessed locally (at the most painful site of the lower back) and remotely (at the contralateral wrist) using the TSA limits protocol:
  * Cold Detection Threshold (CDT)
  * Warmth Detection Threshold (WDT)
  * Cold Pain Threshold (CPT)
  * Heat Pain Threshold (HPT)
Thermal Detection and Pain Threshold Temperatures | FU2 (12 months follow-up)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc Advanced Thermosensory Stimulator (TSA) - 2 system will be used to perform a standardized test protocol.
  Detection and pain threshold temperatures (in °C) will be assessed locally (at the most painful site of the lower back) and remotely (at the contralateral wrist) using the TSA limits protocol:
  * Cold Detection Threshold (CDT)
  * Warmth Detection Threshold (WDT)
  * Cold Pain Threshold (CPT)
  * Heat Pain Threshold (HPT)
Temporal Summation of Pain (TSP) | PRE (baseline)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Temporal summation of pain (TSP) will be assessed at the contralateral wrist using a 2-minute tonic heat stimulus and patient-controlled temperature. Participants are presented with a tonic heat stimulus and are instructed to maintain their initial sensation for two minutes via the remote controller. To quantify temporal adaptation and temporal summation of pain, the slope and magnitude of temperature changes will be extracted and the areas under the curve will be calculated.
Temporal Summation of Pain (TSP) | MID (6 weeks)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Temporal summation of pain (TSP) will be assessed at the contralateral wrist using a 2-minute tonic heat stimulus and patient-controlled temperature. Participants are presented with a tonic heat stimulus and are instructed to maintain their initial sensation for two minutes via the remote controller. To quantify temporal adaptation and temporal summation of pain, the slope and magnitude of temperature changes will be extracted and the areas under the curve will be calculated.
Temporal Summation of Pain (TSP) | POST (12 weeks)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Temporal summation of pain (TSP) will be assessed at the contralateral wrist using a 2-minute tonic heat stimulus and patient-controlled temperature. Participants are presented with a tonic heat stimulus and are instructed to maintain their initial sensation for two minutes via the remote controller. To quantify temporal adaptation and temporal summation of pain, the slope and magnitude of temperature changes will be extracted and the areas under the curve will be calculated.
Temporal Summation of Pain (TSP) | FU1 (3 months follow-up)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Temporal summation of pain (TSP) will be assessed at the contralateral wrist using a 2-minute tonic heat stimulus and patient-controlled temperature. Participants are presented with a tonic heat stimulus and are instructed to maintain their initial sensation for two minutes via the remote controller. To quantify temporal adaptation and temporal summation of pain, the slope and magnitude of temperature changes will be extracted and the areas under the curve will be calculated.
Temporal Summation of Pain (TSP) | FU2 (12 months follow-up)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. QST is a non-invasive examination of the somatosensory system commonly used in pain diagnosis. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Temporal summation of pain (TSP) will be assessed at the contralateral wrist using a 2-minute tonic heat stimulus and patient-controlled temperature. Participants are presented with a tonic heat stimulus and are instructed to maintain their initial sensation for two minutes via the remote controller. To quantify temporal adaptation and temporal summation of pain, the slope and magnitude of temperature changes will be extracted and the areas under the curve will be calculated.
Conditioned Pain Modulation (CPM) | PRE (baseline)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Conditioned pain modulation will be evaluated using a Dual-Thermode program with two different stimuli:
  Test stimulus: this heat stimulus will be administered twice at the contralateral wrist. Once on its own before administering the conditioning stimulus, and once during the conditioning heat stimulus at the ipsilateral wrist.
  Conditioning stimulus: this heat stimulus will be administered at the ipsilateral wrist after first applying the test stimulus.
  The difference in pain intensity at the contralateral wrist during the stand-alone test stimulus and the test stimulus during the conditioning stimulus will be calculated. Pain intensity is assessed using a Numerical Pain Rating Scale (NPRS) ranging from 0 to 100, where 0 stands for "no pain", and 100 for "worst imaginable pain".
Conditioned Pain Modulation (CPM) | MID (6 weeks)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Conditioned pain modulation will be evaluated using a Dual-Thermode program with two different stimuli:
  Test stimulus: this heat stimulus will be administered twice at the contralateral wrist. Once on its own before administering the conditioning stimulus, and once during the conditioning heat stimulus at the ipsilateral wrist.
  Conditioning stimulus: this heat stimulus will be administered at the ipsilateral wrist after first applying the test stimulus.
  The difference in pain intensity at the contralateral wrist during the stand-alone test stimulus and the test stimulus during the conditioning stimulus will be calculated. Pain intensity is assessed using a Numerical Pain Rating Scale (NPRS) ranging from 0 to 100, where 0 stands for "no pain", and 100 for "worst imaginable pain".
Conditioned Pain Modulation (CPM) | POST (12 weeks)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Conditioned pain modulation will be evaluated using a Dual-Thermode program with two different stimuli:
  Test stimulus: this heat stimulus will be administered twice at the contralateral wrist. Once on its own before administering the conditioning stimulus, and once during the conditioning heat stimulus at the ipsilateral wrist.
  Conditioning stimulus: this heat stimulus will be administered at the ipsilateral wrist after first applying the test stimulus.
  The difference in pain intensity at the contralateral wrist during the stand-alone test stimulus and the test stimulus during the conditioning stimulus will be calculated. Pain intensity is assessed using a Numerical Pain Rating Scale (NPRS) ranging from 0 to 100, where 0 stands for "no pain", and 100 for "worst imaginable pain".
Conditioned Pain Modulation (CPM) | FU1 (3 months follow-up)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Conditioned pain modulation will be evaluated using a Dual-Thermode program with two different stimuli:
  Test stimulus: this heat stimulus will be administered twice at the contralateral wrist. Once on its own before administering the conditioning stimulus, and once during the conditioning heat stimulus at the ipsilateral wrist.
  Conditioning stimulus: this heat stimulus will be administered at the ipsilateral wrist after first applying the test stimulus.
  The difference in pain intensity at the contralateral wrist during the stand-alone test stimulus and the test stimulus during the conditioning stimulus will be calculated. Pain intensity is assessed using a Numerical Pain Rating Scale (NPRS) ranging from 0 to 100, where 0 stands for "no pain", and 100 for "worst imaginable pain".
Conditioned Pain Modulation (CPM) | FU2 (12 months follow-up)
  Thermal Quantitative sensory testing (QST) will be used to investigate nociceptive stimulus processing. The Medoc TSA-2 system will be used to perform a standardized test protocol.
  Conditioned pain modulation will be evaluated using a Dual-Thermode program with two different stimuli:
  Test stimulus: this heat stimulus will be administered twice at the contralateral wrist. Once on its own before administering the conditioning stimulus, and once during the conditioning heat stimulus at the ipsilateral wrist.
  Conditioning stimulus: this heat stimulus will be administered at the ipsilateral wrist after first applying the test stimulus.
  The difference in pain intensity at the contralateral wrist during the stand-alone test stimulus and the test stimulus during the conditioning stimulus will be calculated. Pain intensity is assessed using a Numerical Pain Rating Scale (NPRS) ranging from 0 to 100, where 0 stands for "no pain", and 100 for "worst imaginable pain".

CONTACTS AND LOCATIONS:
Overall Officials: Annick Timmermans, Principal Investigator — REVAL-Rehabilitation Research Center, Hasselt University, Diepenbeek, Belgium
Locations (1):
- Hasselt University, Diepenbeek, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No